CLINICAL TRIAL: NCT02727725
Title: Establishing the Clinical Usefulness Of Dark Blood Late Gadolinium Enhancement Images For The Detection Of Small Subendocardial Left Ventricular Infarcts - An Evaluation Of The Novel TRAMINER Sequence By Comparison To Late Gadolinium Enhancement Images
Brief Title: An Evaluation Of The Novel TRAMINER Sequence By Comparison To Late Gadolinium Enhancement Images
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Siemens Corporation, Corporate Technology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AHC IRB 5886
Record Dates: First submitted 2016-02-24; First posted 2016-04-05 (Estimated); Last update posted 2024-10-04 (Actual); Status verified 2018-03

CONDITIONS: Myocardial Fibrosis; Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Traminer MRI Sequence (Experimental): The TRAMINER MRI sequence implementation to be tested allows the acquisition of high resolution MR images in the free-breathing patient, by combining multiple averages and motion correction with the TRAMINER preparation.
  Interventions: Other: Traminer MRI Sequence

INTERVENTIONS:
Other: Traminer MRI Sequence — The Traminer MRI sequence will be added to the standard IR Turbo-Flash sequence and last 2-5 minutes.

SUMMARY:
* The purpose of this study is to show that the novel TRAMINER (T(Rho) and Magnetization Transfer and Inversion Recovery) sequence provides at least as good visualization and detection of sub-endocardial scarring, fibrosis, and acute infarction as the current gold standard Inversion Recovery (IR) Turbo-Flash sequence.
* The hypothesis is that the TRAMINER sequence has the same or higher sensitivity in detecting small sub-endocardial scarring than the inversion recovery segmented gradient echo sequence known as IR-Turbo Fast low angle shot (IR Turbo-Flash), which is the accepted current gold standard for the detection of myocardial viability.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age referred for a cardiac MRI with Gadolinium enhancement only at Advocate Lutheran General Hospital

Exclusion Criteria:

* <18 years old,
* Adults unable to consent
* Adults for whom the MRI has not been previously scheduled
* Adults with an order for any MRI other than cardiac MRI with Gadolinium enhancement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Sensitivity of the TRAMINER sequence in detecting myocardial fibrosis or acute infarction compared to the gold standard sequence will be measured. | 6-12 months
  The method of assessment is through a score using the 17 segment model of myocardial map.

SECONDARY OUTCOMES:
Reduction in clinical Magnetic Resonance (MRI) procedure time. | 6-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Nayla Chaptini, MD, Principal Investigator — Advocate Lutheran General Hospital
Locations (1):
- Advocate Lutheran General Hospital, Park Ridge, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Publication